CLINICAL TRIAL: NCT07055334
Title: Development and Improvement of Home Rehabilitation Scheme for Preschool Children With Congenital Heart Disease After Operation
Status: Not yet recruiting | Type: Observational
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Associate professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: LSLL2024-801
Record Dates: First submitted 2025-06-05; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Heart Defects, Congenital; Rehabilitation; Preschool Child; Qualitative Research; Caregivers; Medical Staff, Hospital
Keywords: congenital heart disease; home-based cardiac rehabilitation; Primary caregiver; qualitative research; preschool child
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This part of the study focuses on understanding the home rehabilitation situation for preschool children with congenital heart disease after operation. Qualitative research interviews with caregivers and medical staff (including doctors, nurses, rehabilitation therapists, nutritionists, and psychologists) are conducted to explore the benefits, obstacles, and professional guidance needs of home rehabilitation. The aim is to summarize the best evidence for home rehabilitation through evidence-based nursing and qualitative research, in order to develop a more comprehensive and suitable home rehabilitation scheme for these children.

ELIGIBILITY:
Children With Congenital Heart Disease After Surgery

Inclusion Criteria:

* Age 3 to 7 years
* Clinical diagnosis of congenital heart disease
* Underwent a single open-heart surgical correction under direct vision at the study site
* Ability to communicate in Chinese

Exclusion Criteria:

* Postoperative arrhythmia
* Comorbid neurological, respiratory, or other systemic diseases
* Deemed unsuitable for exercise by a physician
* Cardiac function classified as NYHA Class IV
* Intellectual, language, or motor impairments resulting from perioperative complications or other causes

Caregivers of Children With Congenital Heart Disease After Surgery

Inclusion Criteria:

* Primary caregiver who voluntarily provides care
* Caregiver who spends the most time with the child
* Ability to communicate in Chinese

Exclusion Criteria:

* Caregivers of children who voluntarily discontinued treatment before completion
* Paid or professional caregivers
* Diagnosed cognitive impairment or mental illness
* Inability to communicate effectively through spoken language
* Presence of serious conflict or instability in the caregiver-child relationship
* Inability to independently operate or use smart electronic devices and the internet

Medical Professionals Involved in Congenital Heart Disease Care

Inclusion Criteria:

* Licensed healthcare professionals, including physicians, nurses, dietitians, physical therapists, or psychological counselors
* At least 5 years of professional experience in congenital heart disease care, rehabilitation, or education

Exclusion Criteria:

* Not currently engaged in frontline clinical work
* Not engaged in clinical work within the past year due to leave, study, or reassignment

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study includes three groups. For children with congenital heart disease after surgery, inclusion criteria are age 3 to 7, one-time corrective open-heart surgery in the research unit, and ability to communicate in Chinese. Exclusions are arrhythmia after surgery, other diseases unsuitable for exercise, heart function class IV, and perioperative disorders.
  For caregivers, must be main caregiver, volunteer, spend most time caring, and communicate in Chinese. Exclusions are those who give up treatment, are paid caregivers, have cognitive impairment or mental illness, cannot express feelings, have contradictions with child, or cannot use electronic devices.
  For medical professionals, must hold license and have at least 5 years of related practice. Exclusions are non-frontline staff or those absent in recent year.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Core Components Finalized in the Home Rehabilitation Scheme Based on Expert Consensus | 12 months (from initiation to completion of scheme development)
  The home rehabilitation scheme will be developed using a two-round Delphi method with a multidisciplinary expert panel. Each proposed module will be rated by experts for its relevance, feasibility, and clarity. Components reaching ≥75% agreement (rated as "agree" or "strongly agree") will be considered finalized. The outcome will be reported as the number and percentage of components finalized out of all proposed components.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Wei, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No